CLINICAL TRIAL: NCT02015403
Title: TO COMPARE THE EFFICACY OF N -ACETYLCYSTEINE AND STANDARD THERAPY VERSUS STANDARD THERAPY IN THE PREVENTION OF ISCHEMIC HEPATITIS AND SURVIVAL POST UPPER GI BLEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-IH-01
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2015-03

CONDITIONS: Ischemic Hepatitis
MeSH Terms: interventions — Standard of Care; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care + NAC (N-ACETYLCYSTEINE) infusion (Experimental)
  Interventions: Drug: Standard Care + NAC (N -ACETYLCYSTEINE); Drug: Standard Care (in control arm)
- Standard Care (Active Comparator)
  Interventions: Drug: Standard Care (in control arm)

INTERVENTIONS:
Drug: Standard Care + NAC (N -ACETYLCYSTEINE)
  Arms: Standard Care + NAC (N-ACETYLCYSTEINE) infusion
Drug: Standard Care (in control arm)

SUMMARY:
Patient presenting with upper GI bleed in ILBS (Institute of Liver and Biliary Sciences) emergency admitted to ICU (Intensive Care Unit) or shifted from ward to ICU (Intensive Care Unit) in view of upper GI bleed randomized to two groups

GROUP A : 110 Patients will receive standard care + NAC infusion for 72 hours

GROUP B : 110 Patients will receive standard care only

NAC will be given at following rate :

Initial loading of 150 mg/kg/hr over 1 hour Followed by 12.5mg/kg/hr for 4 hrs Then continuous infusion of 6.25 mg/kg for the remaining 67 hrs

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 75
* Cirrhotics with UGIE (Upper Gastrointestinal Endoscopy ) within last 24 hours.

Exclusion Criteria:

* Non cirrhotic
* Hepatocellular carcinoma
* Advanced cardiopulmonary disease
* Pregnancy
* Extrahepatic malignancy
* Patient on anticoagulation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To study the efficacy of NAC (N -ACETYLCYSTEINE) in preventing ischemic hepatitis in cirrhotics with upper Gastrointestinal bleed. | Day 5

SECONDARY OUTCOMES:
To study effect of NAC (N -ACETYLCYSTEINE) infusion on 5 day survival post bleed. | 6 weeks
To study incidence of complication like AKI (Acute Kidney Injury), HE(Hepatic Encepahlopathy) and SBP(Spontaneous Bacterial Peritonitis). | day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Maiwall R, Kumar A, Bhadoria AS, Jindal A, Kumar G, Bhardwaj A, Maras JS, Sharma MK, Sharma BC, Sarin SK. Utility of N-acetylcysteine in ischemic hepatitis in cirrhotics with acute variceal bleed: a randomized controlled trial. Hepatol Int. 2020 Jul;14(4):577-586. doi: 10.1007/s12072-020-10013-5. Epub 2020 Feb 11. PMID 32048131